CLINICAL TRIAL: NCT01297595
Title: A Phase 1, Open-Label, Single Dose, Randomized, Cross-Over Relative Bioavailability Study Comparing An Oral Liquid Formulation To A Formulated Capsule Of Crizotinib (PF 02341066) In Healthy Volunteers
Brief Title: Relative Bioavailability Of A Crizotinib Oral Liquid Formulation To Crizotinib Formulated Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A8081019
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Results first posted 2012-02-08 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: relative bioavailability; pharmacokinetics; crizotinib; oral liquid formulation; formulated capsule
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- crizotinib (Experimental)
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — Each subject will receive 250 mg single oral doses of oral liquid formulation and formulated capsule of crizotinib separated by at least 14 days.

SUMMARY:
This study will be an open-label, randomized, 2-period, 2-treatment, 2-sequence, cross-over single-dose study employing administration of two oral formulations of crizotinib (OLF and FC) in the fasted state to healthy adult subjects. Twenty-two (22) subjects will be enrolled to obtain at least 20 evaluable subjects who complete the study. Each subject will receive two treatments (A and B) with a washout period of at least 14 days between each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* 12-lead ECG demonstrating QTc >450 msec or a QRS interval >120 msec at screening. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTc or QRS values should be used to determine the subject's eligibility.
* Pregnant or nursing females; females of childbearing potential, including those with tubal ligation.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormonal replacement therapy must be discontinued 28 days prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle Guidelines described in this protocol.
* Subjects who are investigational site staff members or subjects who are Pfizer employees directly involved in the conduct of the trial.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* A positive serology for Hepatitis B or Hepatitis C.
* Subjects who currently smoke.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081019&StudyName=Relative%20Bioavailability%20Of%20A%20Crizotinib%20Oral%20Liquid%20Formulation%20To%20Crizotinib%20Formulated%20Capsule

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib 250 mg FC First, Then Crizotinib 250 mg OLF: Single oral dose of crizotinib 250 milligram (mg) formulated capsule (FC) in first intervention period; and single oral dose of crizotinib 250 mg oral liquid formulation (OLF) in second intervention period. A washout period of at least 14 days was maintained between each crizotinib dose.
- Crizotinib 250 mg OLF First, Then Crizotinib 250 mg FC: Single oral dose of crizotinib 250 mg OLF in first intervention period; and single oral dose of crizotinib 250 mg FC in second intervention period. A washout period of at least 14 days was maintained between each crizotinib dose.
Period: First Intervention Period
Arm/Group | Crizotinib 250 mg FC First, Then Crizotinib 250 mg OLF | Crizotinib 250 mg OLF First, Then Crizotinib 250 mg FC
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Washout Period (At Least 14 Days)
Arm/Group | Crizotinib 250 mg FC First, Then Crizotinib 250 mg OLF | Crizotinib 250 mg OLF First, Then Crizotinib 250 mg FC
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Crizotinib 250 mg FC First, Then Crizotinib 250 mg OLF | Crizotinib 250 mg OLF First, Then Crizotinib 250 mg FC
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes participants randomized to receive crizotinib 250 mg FC first and crizotinib 250 mg OLF first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time Zero to Infinite Time [AUC (0 - ∞)]
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hours (hrs) post crizotinib dose
Population: Pharmacokinetic (PK) parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Crizotinib 250 mg FC: Single oral dose of crizotinib 250 mg FC [Reference] in either first intervention period or second intervention period.
- Crizotinib 250 mg OLF: Single oral dose of crizotinib 250 mg OLF [Test] in either first intervention period or second intervention period.
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
ng*hr/mL | 2833 (1099) | 2821 (1086)
Statistical Analysis 1: Comparison: Crizotinib 250 mg FC vs Crizotinib 250 mg OLF; Natural log transformed AUC (0 - ∞) of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as a fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals (CIs) for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. This was an estimation study and there was no formal statistical hypothesis; Test type: Superiority or Other; Ratio of Adjusted Means = 99.58, 90% CI 2-sided [91.08 to 108.87]

2. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
hr | 5.00 [2.00 to 6.00] | 5.00 [2.00 to 6.00]

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
ng*hr/mL | 2696 (1073) | 2679 (1069)
Statistical Analysis 1: Comparison: Crizotinib 250 mg FC vs Crizotinib 250 mg OLF; Natural log transformed AUClast of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as a fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. This was an estimation study and there was no formal statistical hypothesis; Test type: Superiority or Other; Ratio of Adjusted Means = 99.35, 90% CI 2-sided [90.51 to 109.07]

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
ng/mL | 121.0 (38.9) | 117.2 (36.1)
Statistical Analysis 1: Comparison: Crizotinib 250 mg FC vs Crizotinib 250 mg OLF; Natural log transformed Cmax of crizotinib was analyzed using a mixed effect model with sequence, period and treatment as a fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. This was an estimation study and there was no formal statistical hypothesis; Test type: Superiority or Other; Ratio of Adjusted Means = 96.84, 90% CI 2-sided [88.22 to 106.32]

5. Secondary Outcome: Plasma Terminal Half-Life (t1/2)
Description: Plasma terminal half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
hr | 35.58 (6.12) | 36.35 (5.64)

6. Secondary Outcome: Apparent Oral Clearance (CL/F)
Description: Drug clearance (CL) is a quantitative measure of the rate at which a drug substance is removed from the plasma. Clearance obtained after oral dose (apparent oral clearance [CL/F]) is influenced by the fraction of the dose absorbed (F).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Liter/hour (L/hr)
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
Liter/hour (L/hr) | 88.21 (30.17) | 88.61 (28.96)

7. Secondary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Liter
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
Liter | 4473 (2089) | 4593 (2108)

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Crizotinib Metabolite (PF-06260182)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast) of Crizotinib metabolite (PF-06260182).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
ng*hr/mL | 429.5 (242.3) | 439.1 (271.5)

9. Secondary Outcome: Area Under the Curve From Time Zero to Infinite Time [AUC (0 - ∞)] for Crizotinib Metabolite (PF-06260182)
Description: AUC (0 - ∞)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞) of crizotinib metabolite (PF-06260182).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: PK parameter analysis population included all participants randomized and treated who had at least 1 of the PK parameters of primary interest in at least 1 treatment period. 'N' = Number of participants contributing to the mean.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 21 | 22
ng*hr/mL | 454.4 (242.1) | 446.7 (273.1)

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
ng/mL | 30.98 (10.39) | 32.56 (10.75)

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Crizotinib Metabolite (PF-06260182)
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
hr | 5.00 [4.00 to 6.00] | 5.00 [4.00 to 6.00]

12. Secondary Outcome: Metabolite to Parent Ratio of Maximum Observed Plasma Concentration (MRCmax)
Description: Metabolite (PF-06260182) to parent (crizotinib) molar ratio of maximum observed plasma concentration (MRCmax).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
Ratio | 0.2482 (0.0349) | 0.2694 (0.0532)

13. Secondary Outcome: Metabolite to Parent Ratio of Area Under the Curve From Time Zero to Last Quantifiable Concentration (MRAUClast)
Description: Molar ratio of metabolite to parent area under the plasma concentration time-curve from time zero (pre-dose) to the last measured concentration (MRAUClast).
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 2
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 22 | 22
Ratio | 0.1546 (0.0275) | 0.1589 (0.0274)

14. Secondary Outcome: Metabolite to Parent Ratio of Area Under the Curve From Time Zero to Infinite Time [MRAUC (0- ∞)]
Description: Molar ratio of metabolite to parent area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0- ∞) [MRAUC (0- ∞)].
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 and 144 hrs post crizotinib dose
Population: as for outcome 9
Measure: Geometric Mean (Standard Deviation); unit: Ratio
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Number analyzed (Participants) | 21 | 22
Ratio | 0.1514 (0.0254) | 0.1535 (0.0259)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Crizotinib 250 mg FC | Crizotinib 250 mg OLF
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 17/22 | 17/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib 250 mg FC (N=22) | Crizotinib 250 mg OLF (N=22)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 6 | 6
Fatigue (General disorders) | 1 | 1
Feeling cold (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 7
Hypersomnia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Abnormal dreams (Psychiatric disorders) | 1 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.